CLINICAL TRIAL: NCT05397951
Title: Evaluation of Wearable Multi-modality Sensors for Monitoring Vital Signs
Brief Title: The Validation Study of Bioelectronics
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 22-0163; 550KR272101 (Other Grant/Funding Number: NC TraCS Pilot Award)
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Healthy; Health Behavior
Keywords: sensor; non-invasive; multi-modality; vital signs; safe wearability; optoelectronic system; optical polarimetry; near-infrared spectroscopy; skin-interfaced; wearable
MeSH Terms: conditions — Health Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- Wearing Biosensor Before & After Exercise (Experimental): Each study participant will wear the bioelectronic sensors during a slow deep breath. Participants will wear the sensors and devices for 15 minutes before and after a brisk 6-minute walk.
  Interventions: Device: Multi-modality Noninvasive Biosensor; Device: Oximeter; Device: Portable Blood Pressure Monitor; Device: Vicorder Pulse Wave Velocity Monitor
- Wearing Biosensor for an Extended Period (Experimental): Each study participant will wear the bioelectronic sensors during a slow deep breath. Participants will wear the sensors and devices continuously for 2 hours.
  Interventions: Device: Multi-modality Noninvasive Biosensor; Device: Oximeter; Device: Portable Blood Pressure Monitor; Device: Vicorder Pulse Wave Velocity Monitor

INTERVENTIONS:
Device: Multi-modality Noninvasive Biosensor — The wearable sensor devices will be placed on the finger, wrist, temple, subclavian, arm, neck, and thigh of the participant and will provide continuous tissue mechanics, heart rate, respiration rate, blood flow, and pulse oxygenation measurements continuously throughout the experimental period.
Device: Oximeter — The oximeter device will be placed on the right middle finger of the participant and will provide continuous pulse oxygenation and heart rate measurements continuously throughout the experimental period.
  Other Names: Abbott Medquip
Device: Portable Blood Pressure Monitor — The blood pressure monitor device will be placed on the left arm of the participant and will take a blood pressure measurement every 5 minutes throughout the 15 minute experimental period, and every 15 minutes throughout the 2 hour experimental period.
  Other Names: Omron
Device: Vicorder Pulse Wave Velocity Monitor — The pulse wave velocity monitor device will be placed on the right side of the neck and the right thigh and will provide measurements continuously throughout the experimental period.

SUMMARY:
The purpose of this study is to investigate the safe wearability and basic functions of the multi-modality sensors fabricated in the PI lab.

DETAILED DESCRIPTION:
Members of this research team have developed innovative, wearable devices capable of being comfortably and continuously worn while recording diverse physiologic measurements. The purpose of this study is to validate the safe wearability and basic functions of the novel biocompatible electronic sensor that will allow continuous, non-invasive physiological measurements. This study aims to obtain preliminary data on the safety and functional aspects of the developed devices and compare it to approved medical equipments (including Abbott Medquip Oximeter, Omron blood pressure monitor, and Vicorder device for pulse wave velocity), which will pave the way for future study that focuses certain disease model. Participants will be randomly assigned to Condition A, and wear the devices before and after exercise for 15 minutes each time, or Condition B and wear the devices for 2 hours continuously. During their 1-hour or 2.5-hour lab visit, study participants will wear the biocompatible electronic sensors and three approved medical devices during a slow deep breath, before and after a 6-minute brisk walk, or for an extended period of time (2 hours). Participants will return to the lab for two brief visits, 48 and 96 hours after the device wearing, to determine if any suspected adverse events related to study procedures or devices emerged after they left the research site. For the future study, we will plan to 1) optimize the devices for use in patients needing FiO2 weaning, 2) demonstrate the reliability, and accuracy of these devices for continuous physiological measurements, including but not limited to blood pressure, heart rate (HR), cerebral blood flow, temperature, glucose concentration, and respiratory rate, and 3) demonstrate these devices are preferred by patients to current measurement tools. Once validated, such sensors could fundamentally change the way blood flow, blood pressure, or related parameters are monitored for patients, eliminating risks associated with invasive monitoring, allowing continuous, real-time detection of clinically meaningful changes in the patients, advancing knowledge of hormonal signatures and physiological signals preceding clinically meaningful events.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with ages between 18 and 99.
* Healthy individuals (not known to suffer any significant illness relevant to the proposed study).

Exclusion Criteria:

* Pregnant or lactating.
* History of active (clinically significant) skin disorders that make skin vulnerable to contact conventional electronic devices.
* History of allergic response to silicones or adhesives (such as 3M Tegaderm).
* Broken, damaged or irritated skin or rashes near the sensor application sites (finger, wrist, temple, subclavian, arm, neck, and thigh).
* Subjects who are physically or cognitively unable to normally perform activities of daily living, assessed at the discretion of the investigator to ensure safe completion of study tasks.
* Subjects who are unable to participate in moderate exercise for 6 minutes.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-01-09 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Mean Comfort Level of Wearable Sensors | Questionnaire completed within 96 hours after device application.
  A questionnaire about the comfort of the wearable sensors will be measured using the Likert scale, which ranges from 1 to 5 and is used to measure attitudes and perception changes about the our sensor. The minimum value 1 represents "strongly disagree" and the maximum value 5 represents "strongly agree", thus higher scores represent a better outcome.
Mean Safety Level of Wearable Sensors | Questionnaire completed within 96 hours after device application.
  A questionnaire about the safety and reactions to the wearable sensors will be measured using the Likert scale, which ranges from 1 to 5 and is used to measure attitudes and perception changes about the safety of our sensor. The minimum value 1 represents "strongly disagree" and the maximum value 5 represents "strongly agree", thus higher scores represent a better outcome.
Mean Agreement Over Time of Physiological Parameters between Newly-Fabricated Wearable Sensors and Approved Devices | Through study completion, an average of 15 minutes.
  Signals from the approved medical devices will measure tissue mechanics, heart rate, respiration rate, blood flow, and pulse oxygenation measurements and these data will be compared to the signals from our sensors. The difference over time will be measured on a scale from a minimum of 0 and a maximum of 1, with 0 being the best outcome and representing the lowest difference between the sensing data from the different devices.

CONTACTS AND LOCATIONS:
Overall Officials: Wubin Bai, PhD, Principal Investigator — Assistant Professor of Applied Physical Sciences
Locations (1):
- Kenan Laboratories at the University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results may be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with the University of North Carolina at Chapel Hill.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 9 and continuing for 36 months following publication.
Access Criteria: Investigator has approved IRB, IEC, or REB and an executed data use/sharing agreement with the University of North Carolina at Chapel Hill.